CLINICAL TRIAL: NCT02099565
Title: Observational Prospective Study to esTIMAte the Rates of Outcomes in Patients Undergoing PCI (Percutaneuos Coronary Intervention) With Drug Eluting Stent (DES) Implantation Who Take Statins (OPTIMA II) - Follow-up
Brief Title: Observational Prospective Study OPTIMA II - Follow-up
Acronym: OPTIMAII
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRU-CRE-2014/1
Record Dates: First submitted 2014-03-25; First posted 2014-03-31 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Major Adverse Cardiovascular and Cerebrovascular Events (MACCE)
Keywords: Major Adverse Cardiovascular and Cerebrovascular Events (MACCE); Statins; LDL-cholesterol; Inflammatory markers; Percutaneous Coronary Intervention (PCI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OPTIMA study patients: The study population will consist of OPTIMA study patients who have not been lost for follow-up and have given a written informed consent.

SUMMARY:
The current follow-up study was planned to reveal the rates of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) during 4-year follow-up in patients participated in OPTIMA study. In addition, the long-term effects of statins on LDL-cholesterol and different biomarkers in patients after drug-eluting stents implantation will be assessed. In addition, such project implementation will allow to clarify the treatment options used by Russian patients with CAD (Coronary Artery Disease) after drug-eluting stent implantation. The information received in this study will help to optimize management of Russian patients with CAD after PCI in order to improve prognosis and quality of life of these patients.

DETAILED DESCRIPTION:
This project is 3-years follow-up of OPTIMA study. This is an observational retro-prospective study based on the data collected during one visit: 4-year after PCI performed at the Russian Cardiological Research Center (РКНПК). From the date of the study start and until the end of the study investigators will enroll those patients participated in OPTIMA study. Only patients, who consent to participate in the study and sign the informed consent form after being informed by a physician on the objectives and methods of the study, will be enrolled into this project.

This study is an observational one, and there is no intervention into routine clinical practice either in terms of therapy, or special examinations. The main point of this project is the data collection using the out-patient medical records or disease history of a patient, as well as collection of data received during patient routine examination. Data collection will be performed only once during single routine patient visit to treating physician or hospitalized patient examination. Study participation will be finished after this visit. Data collection will be performed at the visit 4 years after PCI and will include medical history, current medications, physical examination, ECG (electrocardiogram) and laboratory assessments.

The study will be conducted in Russian Federation. It is planned that 80-90% of patients participated in OPTIMA study will be enrolled into current project. One clinical site - Russian Cardiological Research Center (РКНПК) - is supposed to participate in this study.

The total period of the study is anticipated to be about 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in OPTIMA study;
2. Written informed consent provided prior the start of follow-up in the study

Exclusion Criteria:

1. Lost to follow-up patients of OPTIMA study;
2. Subjects who are unwilling or unable to provide informed consent.

Ages: 18 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Follow-up OPTIMA (NIS-GRU-NEX-2009/) study patients
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The rates of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) in patients after drug-eluting stents (DES) implantation who takes statins at baseline after 4 years after PCI (Percutaneuos Coronary Intervention). | from 1 Jul 2015 to 30 Sep 2015 (after study report preparation)
  The rates of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) in patients after drug-eluting stents (DES) implantation who take statins at baseline after 4 years after PCI.

SECONDARY OUTCOMES:
The proportion of patients who take statins during 4 years after PCI and who discontinue statin therapy. | Up to 4 years after PCI
  The proportion of patients who take statins during 4 years after PCI and who discontinue statin therapy.
The proportion of patients who achieve target level of Low Density Lipoprotein Cholesterol (LDL-C) less than 1,8 mmol/l. | from 1 Jul 2015 to 30 Sep 2015 (after study report preparation)
  The proportion of patients who achieve target level of Low Density Lipoprotein Cholesterol (LDL-C) less than 1,8 mmol/l.
LDL-C level. | from 31 March 2014 to 31 March 2015
  LDL-C level.
Lipoprotein A level. | from 31 March 2014 to 31 March 2015
  Lipoprotein A level.
To estimate adherence to the therapy with statins according to questionnaire based on results of questionnaire | Up to 4 years after PCI
  To estimate adherence to the therapy with statins according to questionnaire based on results of questionnaire
To evaluate proportion of patients who discontinue statin therapy, beta-blockers and ACE (Angiotensin Converting Enzyme) inhibitors therapy and identify their characteristics based on results of questionnaires and CRFs (Case Report Forms) | Up to 4 years after PCI
  To evaluate proportion of patients who discontinue statin therapy, beta-blockers and ACE inhibitors therapy and identify their characteristics based on results of questionnaires and CRFs
To estimate Seattle angina questionnaire (SAQ) score 4 years after PCI | from 1 Jul 2015 to 30 Sep 2015
  To estimate Seattle angina questionnaire (SAQ) score 4 years after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Karin Otter, PHD, MD, Study Director — AstraZeneca; Yuri Karpov, Principal Investigator — Russian Cardiology Research and Production Complex
Locations (1):
- Research Site, Moscow, Russia

REFERENCES:
- [Derived] Karpov Y, Logunova N, Tomilova D, Buza V, Khomitskaya Y. Observational Prospective study to esTIMAte the rates of outcomes in patients undergoing PCI with drug-eluting stent implantation who take statins -follow-up (OPTIMA II). Curr Med Res Opin. 2017 Feb;33(2):253-259. doi: 10.1080/03007995.2016.1253552. Epub 2016 Nov 29. PMID 27779436
- See also: CSR synopsis for OPTIMA II NIS study — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2910&filename=Synopsis.pdf